CLINICAL TRIAL: NCT04682873
Title: A Multi-centre, Double-blind, Randomised, Placebo-controlled, Trial to Assess the Efficacy and Safety of Amizon® Max, Manufactured by Farmak JSC, in Combination With Basic Treatment, in Subjects With Moderate Covid-19, Which is Caused by the SARS-CoV-2 Virus
Brief Title: A Clinical Study to Assess the Efficacy and Safety of Amizon® Max in the Treatment of Moderate Covid-19, Caused by the SARS-CoV-2 Virus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FK/FAV00А-CoV/2020
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Covid-19 Disease
Keywords: Amizon; Antiviral; Covid-19; Enisamium iodide; Ukraine; FAV00A
MeSH Terms: conditions — COVID-19 | interventions — enisamium iodide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Capsule formulations of the placebo Amizon® Max (IMP-2) is identical in appearance (size, shape, and color), taste, and smell as the active drug capsule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enisamium iodide (Experimental): Hospitalized patients who were randomized in to this treatment group will receive enisamium iodide containing capsules (Amizon® Max).
  Interventions: Drug: Enisamium Iodide
- Placebo (Placebo Comparator): Hospitalized patients who were randomized in to this treatment group will receive placebo containing capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enisamium Iodide — Capsule formulations of the active product (enisamium iodide 500 mg; Investigational medicinal product 1 [IMP-1]).
  1 capsule Amizon® Max contains: enisamium iodide 500 mg.
  Amizon® Max (active ingredient: enisamium iodide; IMP-1 will be administered as 1 capsule 4 times a day, every 6 hours (total dose 2,000 mg per day). Capsule will be taken orally (swallowed whole), together with a sufficient amount of liquid (preferably water).
  Treatment will start on Day 1 (randomization) and for up to 168 hours after the first dose administration i.e. Day 7 or Day 8. The site staff will ensure that the IMP (1 capsule) is taken every 6 hours by the study subjects.
  For documentation purposes, the IMP-1 packs (empty blister / blister with unused capsules) will be kept at the site and drug accountability forms are completed.
  Other Names: Amizon, Amizon® Max
  Arms: Enisamium iodide
Drug: Placebo — Capsule formulations of the reference product placebo Amizon® Max (IMP-2), will be identical in appearance (size, shape, and color), taste, and smell as the active formulation capsule.
  1 capsule placebo Amizon® Max contains: placebo (no active substance).
  Amizon® Max placebo (IMP-2), will be administered as 1 capsule 4 times a day every 6 hours. Capsule will be taken orally (swallowed whole), together with a sufficient amount of liquid (preferably water).
  Treatment will start on Day 1 (randomization) and for up to 168 hours after the first dose administration i.e. Day 7 or Day 8. The site staff will ensure that the IMP (1 capsule) is taken every 6 hours by the study subjects.
  For documentation purposes, the IMP-2 packs (empty blister / blister with unused capsules) will be kept at the site and drug accountability forms are completed.
  Arms: Placebo

SUMMARY:
Adult female and male patients, hospitalized with Covid-19 infection (confirmed by reverse transcription polymerase chain reaction [RT-PCR]), will be screened for participation in this prospective, multi-center, double-blind, randomised, placebo-controlled trial.

Enrolled patients will be randomized (1:1) into 2 treatment groups: Group 1 will receive the active treatment with Amizon® Max (international nonproprietary name enisamium iodide), one capsule (each containing 500 mg of enisamium iodide) 4 times daily every 6 hours for 7 days; patients in treatment Group 2 will receive a matching placebo capsule, 4 times daily every 6 hours for 7 days. Patient observation and follow-up are planned for 29 days, unless discharged before Day 29.

The effect of treatment on Covid-19 will be evaluated by time from day of randomization to an increase of at least two points (from the status at randomization) on the severity rating scale (SR), the Time to Clinical Recovery (TTCR) of main Covid-19 symptoms / complications and the Sum of Severity Rating from Day 2 to Day 15 (SSR-15). Safety and tolerability of the study drug will be evaluated based on the intensity and course of adverse events (Es).

Enisamium iodide is an antiviral small molecule. Enisamium inhibits replication of alpha- and beta- coronaviruses (human coronavirus NL63 and SARS-CoV-2, respectively) and influenza virus A and B. Mechanism of action against SARS-CoV-2 includes the direct inhibition of the viral RNA polymerase.

DETAILED DESCRIPTION:
This randomized, prospective, multi-center, double-blind, placebo-controlled trial, is conducted to investigate the clinical efficacy and safety of the drug Amizon® Max (N-methyl-4-benzylcarbamidopyridinium iodide, international nonproprietary name enisamium iodide, lab code FAV00A) in comparison with placebo, for the treatment of hospitalized patients with RT-PCR confirmed Covid-19 infection.

Enisamium iodide is an antiviral small molecule. Enisamium can directly inhibit influenza viral RNA replication and has antiviral effect against viruses, including coronaviruses (human coronavirus NL63, SARS-CoV-2).Based on the promising in-vitro anti-SARS-CoV-2 activity, it could be assumed that patients suffering from Covid-19 would benefit from a reduced virus load and this could lead to a reduction of Covid-19 typical symptoms that might prevent further complications associated with severe Covid-19 (e.g. active mechanical ventilation).

Adult female and male patients, with Covid-19 infection, will be screened (Day 1) to participate in this trial. If all inclusion/exclusion criteria are fulfilled, randomization to treatment and a start of treatment will occur on Day 1.

Patients will be randomized into 2 treatment groups (1:1) as follows: patients in treatment Group 1 will receive the active treatment with Amizon® Max capsule; patients in treatment Group 2 will receive a placebo capsule. The active treatment and placebo capsules are identical in appearance and size.

Patients will take Amizon® Max capsules 500 mg (active ingredient enisamium iodide) 4 times a day every 6 hours (total daily dose 2,000 mg) for full 7 days. In the control group, patients will take placebo tablets 4 times a day for full 7 days. Patient observation interval is for as long as a subject is hospitalized Day 1 to Day 29. A follow-up visit will be performed on Day 29 (by phone as applicable for all subjects discharged from the hospital before Day 29).

The effect of treatment on Covid-19 will be evaluated by the time from the day of randomization (Day 0) to an improvement of at least two points (from the status at randomization) on the severity rating scale (SR), the Time to Clinical Recovery (TTCR) of main Covid-19 symptoms / complications and the Sum of Severity Rating from Day 2 to Day 15 (SSR-15).

Additional outcome measures of efficacy include the 'Days Alive' and 'Out of Hospital' from Day 1 until Day 15 (DAOH-14), the proportion of subjects discharged by Day 8, 15, 22, and 29, the incidence of complications (i.e. pneumonia, need for transfer to intensive care unit [ICU]), the incidence and days until occurrence of pneumonia, incidence and days until supplemental oxygen / high flow oxygen, incidence and days until (non-invasive / invasive mechanical ventilation), incidence and days until transfer to ICU, incidence and time to death, time to virus free, measurement of vital signs (i.e. fever (body temperature), respiratory rate, peripheral capillary oxygen saturation [SpO2]) and the course of symptoms of Covid-19.

Symptom severity for headache, sore throat, cough, shortness of breath, rhinorrhoea, fatigue, myalgia, diarrhoea will be monitored. Safety and tolerability of the study drug will be evaluated based on the intensity and course of adverse events (AEs), safety laboratory tests, as well as the investigator's and subject's overall assessment of tolerability of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be randomized to treatment:

1. Willing and able to provide written informed consent
2. Aged ≥ 18 years
3. SARS-CoV-2 infection confirmed by PCR ≤ 4 days before randomization
4. Currently hospitalized due to SARS-CoV-2 infection with fever, defined as body temperature ≥ 37.8 °C
5. Modified World Health Organization (WHO) Ordinal Scale for Clinical Status Patient state in Covid-19: score 4 i.e. hospitalized, virus-positive, oxygen by mask or nasal prongs

Exclusion Criteria:

The subject is excluded from the trial if any of the following criteria apply:

1. Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 is prohibited < 24 hours prior to start of IMP treatment
2. Requiring mechanical ventilation at screening or it is expected within 24 h after inclusion
3. Expected survival time < 72 hours for any reason
4. Positive pregnancy test
5. Breastfeeding woman
6. Presence of renal dysfunction defined as estimated glomerular filtration rate (eGFR) <60 mL/min, total bilirubin ≥ 2.0 mg/dL, Thyroid stimulating hormone (TSH) outside normal range and / or Aspartate aminotransferase (ASAT)/ Alanine aminotransferase (ALAT) above threefold upper limit of normal range (known from patients medical history)
7. Known hypersensitivity to the trial drug, the metabolites, or formulation excipient
8. History or presence of drug or alcohol abuse
9. History or presence of diseases of thyroid gland

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Efficacy - Time from day of randomization to an improvement of at least two points (from the status at randomization) on severity rating (SR) scale in days | Day 0 to Day 29
  Time from day of randomization to an increase of at least two points (from the status at randomization) on the following severity rating (SR) scale in days:
  1. - Death
  2. - Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. - Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. - Hospitalized, requiring supplemental oxygen
  5. - Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Covid-19 related or otherwise)
  6. - Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. - Not hospitalized, limitation on activities and/or requiring home oxygen
  8. - Not hospitalized, no limitations on activities

SECONDARY OUTCOMES:
Efficacy - Time to recovery (TTR) from Day 1 (randomization and start of IMP treatment) | Day 0 to Day 29
  Time to recovery (TTR) from day of randomisation: Day of recovery is defined as the first day on which the subject satisfies one of the following 3 categories from the ordinal scale (same scale being used as for the primary endpoint):
  6 - Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care 7 - Not hospitalized, limitation on activities and/or requiring home oxygen 8 - Not hospitalized, no limitations on activities
Time to Clinical Recovery (TTCR) of main Covid-19 symptoms/complications or discharge | Day 0 to Day 29
  Time to Clinical Recovery (TTCR) of main Covid-19 symptoms/complications or discharge, whichever comes first: TTCR is defined as the time (Days) from randomisation (active or placebo) until normalization of fever, respiratory rate, oxygen saturation, and cough, sustained for at least 48 hours. Normalization and alleviation criteria:
  * Fever ≤37.2°C
  * Respiratory rate - ≤24/minute on room air
  * Oxygen saturation - >94% on room air
  * Cough: absent
Sum of Severity Rating from Day 2 to Day 15 (SSR-15) | Day 2 to Day 15
  Sum of Severity Rating from Day 2 to Day 15 (SSR-15): Daily reporting of severity rating on an 8-point ordinal scale. The ordinal scale is an assessment of the clinical status starting from initiation of study treatment (active or placebo) from Day 2 to Day 15. The scale from 1 to 8 as defined for the primary endpoint.
Severity Rating on Day 15 (SR-15): | Day 15 or Day of discharge (whichever occurs first)
  Severity Rating on Day 15 (SR-15): Reporting of severity rating on Day 15 or Day of discharge whichever occurs first on an 8-point ordinal scale. The ordinal scale is an assessment of the clinical status. The scale is defined from 1 (Death) to 8 (Not hospitalized, no limitations on activities) as defined for the primary endpoint.
Days Alive and Out of Hospital until Day 15 (DAOH-14) | Day 2 to Day 15
  The number of days alive and discharged from hospital until day 15 will be calculated for each group and the treatment differences displayed.
Proportion of Subjects Discharged by Day 8, 15, 22, 29 | Day 0 to Day 29
  The proportion of subjects discharged by Day 8, 15, 22 and 29 will be displayed for the two treatment groups.
Incidence of non-invasive ventilation | Day 0 to Day 29
  The analysis of the incidences of non-invasive ventilation will be performed by logistic regression model with the binary outcome as dependent variable, age as covariate, baseline severity rating, centre, treatment and centre x treatment as factors.
Days until non-invasive ventilation | Day 0 to Day 29
  The days until non-invasive ventilation will be calculated and the treatment differences displayed using the stratified log-rank test.
Total days of non-invasive ventilation | Day 0 to Day 29
  The total days of non-invasive ventilation will be evaluated by the generalized linear model based on the Poisson distribution and including age as covariate, baseline severity rating, centre, treatment and centre x treatment as factors into the model.
Incidence of invasive mechanical ventilation or ECMO | Day 0 to Day 29
  The analysis of the incidence rate of invasive mechanical ventilation will be performed by logistic regression model with the binary outcome as dependent variable, age as covariate, baseline severity rating, centre, treatment and centre x treatment as factors.
Days until invasive mechanical ventilation or ECMO | Day 0 to Day 29
  The days until invasive mechanical ventilation or ECMO will be calculated and the treatment differences displayed using the stratified log-rank test.
Course of qualitative RT-PCR viral test results | Day 0 to Day 29
  The course of qualitative RT-PCR virus test results will be evaluated by logistic regression with virus test as dependent variable, age as covariate, baseline severity rating, day, centre, treatment as fixed factors. In addition the interaction terms treatment x day and treatment x centre will be included as interaction term as fixed effect into the model. The treatment x day interaction term should detect any differences between treatments in the time until virus deletion.
Viral test evaluation - Proportion of subjects free of SARS-CoV-2 | Days 0, 8, 15, 22, 29
  Proportion of subjects SARS-CoV-2 free pharyngeal swabs / sputum samples (virus-free) on Days 8, 15, 22, 29
Overall assessment of efficacy (patient and investigator) | Day 29 or Day of discharge (whichever occurs first)
  The investigator and the subject (each separately) will assess the overall (global) efficacy of the IMP, based on the change in symptoms using a Four-point verbal rating scale (VRS-4) (0=no symptoms / cured, 1=symptoms improved compared to Visit 1, 2=symptoms unchanged compared to Visit 1, 3=symptoms deteriorated compared to Visit 1).
Adverse events (AEs) | Day 0 to Day 29
  Evaluate AEs by time of onset, actions taken, pattern of occurrence, and outcome
Overall assessment of tolerability of treatment (patient and investigator) | Day 29 or Day of discharge (whichever occurs first)
  Difference in the global tolerability judgement scores on Day of Discharge from hospital (or Day 29, end of trial, if not discharged earlier).
  The investigator and the subject (each separately) will assess the overall (global) tolerability of the IMP using a five-point rating scale (0=very good, 1=good, 2=moderate, 3=poor, 4=very poor).

CONTACTS AND LOCATIONS:
Overall Officials: Olha Holubovska, MD, DSc, Principal Investigator — Head of Department of Infectious Diseases; O.O. Bogomolets National Medical University; Kyiv Ukraine
Locations (13):
- Ukraine (13):
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council, Dept. Pulmonology, Lutsk, Volynsk
  - Municipal Non-Commercial Enterprise 'City Clinical Hospital #3' Chernivtsi City Council, Dept. Therapeutics #1, Dept. Therapeutics #2, Higher State Educational Institution of Ukraine 'Bukovinian State University', Chernivtsi
  - Municipal Non-Commercial Enterprise 'Regional Clinical Infection Hospital Ivano-Frankivsk Regional Council', Dept. #2, Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Municipal Non-Commercial Enterprise 'Regional Clinical Hospital Ivano-Frankivsk Regional Council', Dept. Allergology, Ivano-Frankivsk
  - Municipal Non-Commercial Enterprise 'City Clinical Hospital #1 Ivano-Frankivsk City Council', Dept. Therapeutics, Ivano-Frankivsk
  - Municipal Non-Commercial Enterprise Kharkiv Regional Council 'Regional Clinical Infection Hospital', 1st Department, Kharkiv National Medical University, Chair of Infectious Diseases, Kharkiv
  - Municipal Non-Commercial Enterprise 'Olexandrivska Clinical Hospital of Kyiv' Executive Authority of Kyiv City Council, Dept. Infections, Kyiv
  - Municipal Non-Commercial Enterprise "Kyiv City Clinical Hospital #9" Executive Authority of Kyiv City Council, Dept. Infections, Kyiv
  - Municipal Non-Commercial Enterprise Lviv Regional Council 'Lviv Regional Infection Hospital', Fourth Diagnostic Department, Lviv
  - Ukraine Medical Stomatological Academy, Chair of Infectious Diseases with Epidemiology, Municipal Non-Commercial Enterprise 'Poltava Regional Infection Hospital Poltava Regional Council', Dept. Respiratory Infections, Poltava
  - Municipal Non-Commercial Enterprise 'Central Clinical Hospital' of Rivne City Council, Hepatic Centre - Infections, Rivne
  - Municipal Non-Commercial Enterprise 'Regional Clinical Infectional Hospital' Transcarpathian Regional Council, Dept. Infections (Adult), Uzhhorod
  - Municipal Non-Сommercial Enterprise 'Vinnytsya City Clinical Hospital #1', Infectious Department, National Pirogov Memorial Medical University, Dept. Infections, Vinnytsia

IPD SHARING:
Plan to Share IPD: No